CLINICAL TRIAL: NCT00184613
Title: An Open-label, Randomised, In-patient, Cross Over PK/PD Trial Investigating the Pharmackinectic and Pharmacodynamic Profiles Following Continuous Subcutaneous Infusion of Insulin Aspart or Injection of Insulin Glargine in Subjects With Type 2 Diabetes Mellitus
Brief Title: Comparison of Insulin Glargine Against Insulin Aspart Infused Under the Skin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDS253-1666; 2005-000268-22 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pump
Drug: insulin glargine
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe. The objective of the study is to investigate the effect and safety of continously basal delivered insulin aspart given by a pump versus once daily injection of insulin glargine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes for more than 2 years
* Subjects currently treated with unchanged insulin glargine dose (10 -100 units) for 2 weeks
* Subjects currently treated with unchanged dose(s) for at least 1 month on one or two Oral Anti-diabetic drugs
* BMI 25 - 40 kg/m2
* HbA1c < 9.5 %

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Previous randomisation in this trial
* Pregnancy, breast-feeding, intention of becoming pregnant or pre-menopausal women judged not to be using adequate contraceptive measures (Only sterilisation, intra uterine devices and contraceptive pills are considered adequate contraceptive methods)
* Mental incapacity, unwillingness or language barriers precluding adequate understanding and co-operation.
* Any other significant illness such as endocrine, cardiac, neurological, malignant or other pancreatic illness judged by Investigator
* Participation in other studies within the last three months

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-05; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Variation in morning FPG | Collected in hospital on the last 5 days of 7 days hospitalization, and on the morning of discharge

SECONDARY OUTCOMES:
Variation of plasma endogenous insulin and insulin aspart/glargine collected in hospital on the last 5 days and the morning on discharged
Variation of pre-dinner plasma glucose collected in hospital on the last 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Århus C, Denmark

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com